CLINICAL TRIAL: NCT05395000
Title: Comparison of Ease of Use and Acceptability of Intranasal and Injectable Glucagon Among Providers Administering it to Children or Adolescents With Type 1 Diabetes
Brief Title: Comparison of Ease of Use and Acceptability of Intranasal and Injectable Glucagon Among Providers Administering it to Children or Adolescents With Type 1 Diabetes (BETTER-ING)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Claudia Gagnon, Principal Investigator, Endocrinologist, Regular Researcher of the Endocrinology-Nephrology Axis, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-5626
Record Dates: First submitted 2022-04-29; First posted 2022-05-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia
Keywords: injectable glucagon; intranasal glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Videotape Recording; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Half of the participants will perform the simulation study with the intranasal device first and the other half with the injectable glucagon to minimize the bias related to the lower stress of the second simulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Parents" group (Experimental): Parent or primary caregiver of a child or adolescent (<18 years old) diagnosed with type 1 diabetes.
  Interventions: Behavioral: Videos; Behavioral: Simulation; Behavioral: Interview
- "School workers" group (Experimental): Any adult who works or will work in a school or daycare setting who is likely to administer glucagon to a child or adolescent with type 1 diabetes (e.g. teachers, facilitators, teacher candidates, etc.). This individual must not meet the criteria for the "parent" group.
  Interventions: Behavioral: Videos; Behavioral: Simulation; Behavioral: Interview

INTERVENTIONS:
Behavioral: Videos — A short video explaining briefly what type 1 diabetes is, the symptoms of hypoglycemia and the usefulness of glucagon as well as two short videos explaining how to administer glucagon, all less than 3 minutes long, will be viewed by the 2 groups for intranasal glucagon and injectable glucagon. Participants will have access to the videos for 2 weeks, approximately 3 months before the next stages of the project.
Behavioral: Simulation — An intranasal and injectable glucagon administration test on a mannequin in a simulated stress environment will be done.
Behavioral: Interview — At the end of the simulation, participants will participate in a semi-structured, recorded individual interview of approximately 20 minutes to share their experience related to preferences, barriers, emotional impact, and method of teaching the use of the two glucagon formulations.

SUMMARY:
Background : The benefits of good glycemic control are clearly established. However, achieving glycemic targets comes at the expense of the risk of hypoglycemia. Repeated episodes of severe hypoglycemia can affect long-term cognitive function, especially in developing brains. Fear of hypoglycemia, both in children and their parents, has an impact on participation in physical activity, quality of life and optimal diabetes control. During an episode of severe hypoglycemia, i.e., when accompanied by severe cognitive dysfunction requiring assistance from others, it is impossible to administer oral glucose. Glucagon administration is particularly useful in this situation, as it rapidly raises blood glucose levels and restores consciousness. Injectable glucagon was the only form approved in Canada prior to 2019. A new formulation of glucagon for intranasal administration has recently been approved by Health Canada. The arrival of this formulation seems promising because of its ease of use while ensuring similar efficacy to injectable glucagon. Furthermore, the ease of learning how to use each of the devices through a simple multimedia tool is unknown. Indeed, current studies have not focused on a virtual teaching method. The latter is of particular interest in the context of a pandemic and in order to make information more accessible to a broader population that may not be present at family glucagon education (e.g., school-based caregivers).

Objective : Compare the performance (time to prepare and administer, success rate) of the intranasal versus injectable glucagon administration procedure after a short video training 3 months earlier among parents/primary caregivers and school workers who may administer glucagon to children with type 1 diabetes.

Secondary objectives :

1. To assess stakeholder administration procedure preferences for the two glucagon formulations in the two groups ;
2. To explore the barriers and emotional impact (fears, perceptions, stress, etc.) related to the use of intranasal and injectable glucagon in both groups;
3. Explore the participants' preferences in relation to the teaching method of administering the two forms of glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Parent or primary caregiver of a child or adolescent (<18 years old) diagnosed with type 1 diabetes OR
* Any adult who works or will work in a school or daycare setting who is likely to administer glucagon to a child or adolescent with type 1 diabetes (e.g. teachers, animators, teacher candidates, etc.) AND
* Legal age
* Able to participate

Exclusion Criteria:

* Working in the health field and teach glucagon injection or use it regularly in their duties
* Not understanding French (for viewing the videos)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Time to complete preparation and administration of the glucagon | through the simulation completion, 3 months after listening to the videos
  As an indicator to compare the performance of the intranasal glucagon and injectable glucagon procedures
Success rate of glucagon administration | through the simulation completion, 3 months after listening to the videos
  As an indicator to compare the performance of the intranasal glucagon and injectable glucagon procedures.
  Success is defined as completion of at least 80% of the key steps, including 100% of the "critical" steps

SECONDARY OUTCOMES:
Preferences of the administration procedure for the two glucagon formulations in the two groups | through the interview completion, 3 months after listening to the videos
Barriers related to the use of intranasal and injectable glucagon in both groups | through the interview completion, 3 months after listening to the videos
  The barriers and emotional impact raised by the participants will be classified using the theoretical domains framework (TDF), which is a validated theoretical framework composed of 14 modifiable domains that allows for the assessment of barriers to the implementation of a behavior change and facilitates the development of solution paths afterwards
Emotional impact (fears, perceptions, stress, etc.) related to the use of intranasal and injectable glucagon in both groups | through the interview completion, 3 months after listening to the videos
  The barriers and emotional impact raised by the participants will be classified using the theoretical domains framework (TDF), which is a validated theoretical framework composed of 14 modifiable domains that allows for the assessment of barriers to the implementation of a behavior change and facilitates the development of solution paths afterwards
Preferences in relation to the teaching method of administering the two forms of glucagon | through the interview completion, 3 months after listening to the videos

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, Dr, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- Centre de recherche du CHU de Québec - Université Laval, Québec, Canada

REFERENCES:
- [Derived] Wang YP, Bernatchez F, Chouinard-Castonguay S, Tremblay MC, Vanasse A, Kinnard N, Megalli M, Millette M, Boulet G, Henderson M, Simoneau-Roy J, Brazeau AS, Rabasa-Lhoret R, Gagnon C. Comparison of Intranasal and Injectable Glucagon Administration Among Pediatric Population Responders. Diabetes Technol Ther. 2023 Nov;25(11):808-816. doi: 10.1089/dia.2023.0290. PMID 37751153